CLINICAL TRIAL: NCT06175572
Title: The Diagnostic and Prognostic Value of Comprehensive Functional Assessments for Non-obstructive Coronary Artery Diseases.
Brief Title: Comprehensive Functional Assessments for NOCAD
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Junbo Ge, Professor, Shanghai Zhongshan Hospital
Other Study IDs: ZS20231202
Record Dates: First submitted 2023-12-04; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Coronary Microvascular Dysfunction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- NCF cohort: Normanl coronary-flow patients referred to coronary angiography and undergo assessment with single photon emission computed tomography imaging (SPECT).
  Interventions: Device: coronary physiological indices
- CSF cohort: Coronary slow-flow patients referred to coronary angiography and undergo assessment with single photon emission computed tomography imaging (SPECT).
  Interventions: Device: coronary physiological indices
- ANOCA cohort: Angina with nonobstructive coronary artery patients referred to coronary angiography and undergo assessment with single photon emission computed tomography imaging (SPECT).
  Interventions: Device: coronary physiological indices
- INOCA cohort: Ischemia with nonobstructive coronary artery patients referred to coronary angiography and undergo assessment with single photon emission computed tomography imaging (SPECT).
  Interventions: Device: coronary physiological indices

INTERVENTIONS:
Device: coronary physiological indices — coronary physiological indices

SUMMARY:
To validate and investigate the efficacy of comprehensive functional assessments for the diagnostic and prognostic value in NOCAD.

ELIGIBILITY:
Inclusion Criteria:

1. visual evaluation of epicardial coronary artery diameter stenosis (DS%) ≤ 50%;
2. CZT-SPECT was successfully conducted within three days of CAG

Exclusion Criteria:

1. had flow-limiting epicardial stenosis (DS% >50%) or angiography-derived FFR (Angio-FFR) ≤ 0.8;
2. severe valvular heart disease;
3. chronic heart failure and/or left ventricular ejection fraction (LVEF) of < 50%;
4. cardiomyopathy and myocarditis;
5. severe renal or hepatic insufficiency;
6. failure in detecting SPECT;
7. failure in computing Angio-IMR, and -FFR.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population enrolled from Zhongshan Hospital, Fudan University (Shanghai, China)，with coronary angiography and available cadmium zinc telluride - single photon emission computed tomography imaging (CZT-SPECT).
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | 5 years
  The composite of coronary heart disease death, nonfatal myocardial infarction, hospitalization for unstable angina, or fatal or nonfatal ischemic stroke.

SECONDARY OUTCOMES:
Individual components of MACE | 5 years
  Cumulative incidence of the individual components of MACE
the change in Seattle Angina Questionnaire (SAQ) summary score | 5 years
  The SAQ comprises 5 components namely physical limitation, angina stability, angina frequency, treatment satisfaction, and quality of life; these are then incorporated into the summary score. The higher the score, the better the patient's quality of life and physical function.
the change in Seattle Angina Questionnaire (SAQ) score of indivadual scale | 5 years
  The SAQ comprises 5 components namely physical limitation, angina stability, angina frequency, treatment satisfaction, and quality of life. The higher the score, the better the patient's quality of life or physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Chenguang Li, Study Director — Fudan University
Locations (1):
- Zhongshan hospital, Fudan university, Shanghai, China

IPD SHARING:
Plan to Share IPD: No